CLINICAL TRIAL: NCT07217418
Title: Music Therapy and Its Effects on Premenstrual Syndrome (PMS)
Acronym: PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Chester University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PMSMT2025
Record Dates: First submitted 2025-09-26; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Premenstrual Syndrome; Menstrual Symptoms
Keywords: Music therapy; PMS; Premenstrual syndrome; Music Based Intervention
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Listening Group (Active Comparator)
  Interventions: Behavioral: Music Listening Group (LG)
- Singing Group (Experimental)
  Interventions: Behavioral: Participant-Selected Songs for the Interactive Singing Intervention Group (SG)
- Instrumental Playing Group (Experimental)
  Interventions: Behavioral: Participant-Selected Songs for the Interactive Instrumental Playing Group (PG)

INTERVENTIONS:
Behavioral: Music Listening Group (LG) — The Listening Group (LG) listened to a randomly selected song that featured a slow tempo, a major key, and sedative music, and listened to pre-recorded music for 15-20 minutes without an interventionist. All sessions were conducted individually in a quiet, private music therapy room to ensure a controlled, distraction-free environment. Participants were seated comfortably, and a researcher responsible for monitoring their physiological responses remained present but positioned to avoid direct eye contact.
  Arms: Music Listening Group
Behavioral: Participant-Selected Songs for the Interactive Singing Intervention Group (SG) — The researchers curated a list of 23 songs based on participants' preferred genres and artists, as identified through an initial survey. These songs, characterized by an upbeat tempo (80-110 BPM) and major key tonality, were selected to reflect common musical elements aligned with participants' preferences. All sessions were conducted individually in a quiet, private music therapy room to ensure a controlled, distraction-free environment. Participants were seated comfortably facing the interventionist, while a researcher responsible for monitoring physiological responses remained present but positioned to avoid direct eye contact. Participants in the Singing Group (SG) selected a song from the curated list, received a lyric sheet, and sang along as the interventionist provided vocal and guitar accompaniment.
  Arms: Singing Group
Behavioral: Participant-Selected Songs for the Interactive Instrumental Playing Group (PG) — The researchers selected 23 songs based on participants' preferred genres and artists, as identified through an initial survey. These songs, characterized by an upbeat tempo (80-110 BPM) and major key tonality, were chosen to reflect musical elements commonly found in participants' preferences. All sessions were conducted individually in a quiet, private music therapy room to ensure a controlled, distraction-free environment. Each participant was seated in a comfortable chair facing the interventionist, while a researcher monitoring physiological responses remained present but positioned to avoid direct eye contact. Participants in the Playing Group (PG) selected a preferred song from the curated list and played a full-sized djembe while listening to live music performed by the interventionist, who provided vocal and guitar accompaniment. To maintain rhythmic focus, participants were instructed not to sing while playing the drum.
  Arms: Instrumental Playing Group

SUMMARY:
The purpose of the research is to explore the effects of music therapy on premenstrual syndrome and its symptoms. The goal of this study is to answer the following research questions:

1. Will the passive music listening group and music therapy group (singing and instrumental playing) have a different effect on the physiological responses (EMG, skin conductance, and heart rate) of college students with PMS?
2. Will the passive music listening group and music therapy group (singing and instrumental playing) have a different effect on the brain wave (EEG) of college students with PMS?
3. Will the passive music listening group and music therapy group (singing and instrumental playing) have a different effect on the anxiety level of college students with PMS?
4. Will the passive music listening group and music therapy group (singing and instrumental playing) have a different effect on the pain perception of college students with PMS?
5. How do college students with PMS respond after listening to music, singing, and instrumental playing?

Participants were randomly assigned to one of three groups: a passive music-listening group, an active singing group, or an active instrumental-playing group. Physiological responses were collected before, during, and after the intervention. Participants who volunteered completed a written survey following the intervention.

DETAILED DESCRIPTION:
Upon IRB approval for this research, an email invitation was distributed to a private university in Northeastern Pennsylvania. The Premenstrual Syndrome Scale (PMSS) was used to screen participants to measure the severity of PMS symptoms. PMSS consists of 44 items and has nine sub-dimensions: depressive sensation, anxiety, fatigue, nervousness, depressive thoughts, pain, appetite changes, and sleep pattern. Each item is scored, and a high score indicates intense PMS symptoms. Demographic questions were followed to identify participants' background information, including their musical background, age, and general symptoms of PMS. Once participants were recruited, they were randomly assigned into three groups. The participants in the listening group listened to 30 minutes of meditative music, while the playing and singing groups utilized 30 minutes of either the listening or singing of preferred music led by a music therapy student under a certified music therapist's supervision. Each participant scheduled an appointment with a student music therapist within ten days of their menstrual period. This experiment will consist of several pre-, during, and post-tests. First, participants received an electroencephalogram (EEG) test to measure the electrical activities in their brains through the Biofeedback ProComp Infinity System with BioGraph Infiniti Software-T7500M. Electromyography (EMG) was used to measure the electrical activity of the participant's muscle tension using this equipment. In addition, respiratory rate, heart rate, and temperature were measured. Additionally, the participants completed both an anxiety self-report (State-Trait Anxiety Inventory) and a pain perception self-report pre-and post-test. Finally, 10 participant completed a qualitative questionnaire survey only for their post-test.

ELIGIBILITY:
Inclusion Criteria:

* Participants were biologically female individuals who reported experiencing premenstrual syndrome (PMS) in the initial survey and were currently in their menstrual cycle. Only those who were 7-10 days prior to the onset of their period were eligible to participate in the intervention.

Exclusion Criteria:

* Individuals who identify as transgender women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Alpha Wave Activity (EEG) | It was a one-time intervention on the same day (day 1), each participant with assessments immediately before the intervention (baseline), during the intervention, and immediately after the intervention (post-test).
  Alpha wave activity was measured using electroencephalography (EEG) via the Biofeedback ProComp Infinity System BioGraph Infiniti Software (T7500M). Alpha amplitude was reported in microvolts (µV) to assess relaxation-related brain activity.
Muscle Tension (EMG) | It was a one-time intervention on the same day (day 1), each participant with assessments immediately before the intervention (baseline), during the intervention, and immediately after the intervention (post-test).
  Muscle tension was assessed using electromyography (EMG) recorded with the Biofeedback ProComp Infinity System BioGraph Infiniti Software (T7500M). EMG amplitude was reported in microvolts (µV).
Heart Rate | It was a one-time intervention on the same day (day 1), each participant with assessments immediately before the intervention (baseline), during the intervention, and immediately after the intervention (post-test)
  Heart rate was recorded using the Biofeedback ProComp Infinity System BioGraph Infiniti Software (T7500M) and reported in beats per minute (bpm).
Skin Conductance (SC) | It was a one-time intervention on the same day (day 1), each participant with assessments immediately before the intervention (baseline), during the intervention, and immediately after the intervention (post-test).
  Skin conductance(SC) was recorded using the Biofeedback ProComp Infinity System BioGraph Infiniti Software (T7500M) to evaluate autonomic arousal. Data was expressed in microsiemens (µS).
Anxiety (State-Trait Anxiety Inventory; STAI) | This was a one-time intervention conducted on Day 1. Each participant completed assessments at baseline (pre-intervention, prior to physiological measurements) and immediately post-intervention (following completion of physiological measurements).
  Anxiety levels were assessed using the State-Trait Anxiety Inventory. Scores were reported as units on a scale from 20 to 80, with higher scores indicating greater anxiety.
Pain Perception | This was a one-time intervention conducted on Day 1. Each participant completed assessments at baseline (pre-intervention, prior to physiological measurements) and immediately post-intervention (following completion of physiological measurements).
  Pain perception was measured using a self-report questionnaire. Scores were reported on a numeric rating scale from 0 to 10, with higher scores indicating greater perceived pain intensity.

SECONDARY OUTCOMES:
Qualitative questionnaire survey | Assessments were conducted immediately post-intervention (following completion of physiological, anxiety, and pain measurements). It was a one-time intervention conducted on Day 1.
  A qualitative questionnaire was developed by the investigators and administered only during the post-test. The questionnaire included open-ended questions such as, 'What was your most memorable experience during this live music session?' and 'How did you feel before and after participating in the music-based intervention?

CONTACTS AND LOCATIONS:
Overall Officials: Eun Sil Suh, PhD, Principal Investigator — West Chester University
Locations (1):
- Marywood University, Scranton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saglam HY, Basar F. The relationship between premenstrual syndrome and anger. Pak J Med Sci. 2019 Mar-Apr;35(2):515-520. doi: 10.12669/pjms.35.2.232. PMID 31086543
- [Background] Arjmand HA, Hohagen J, Paton B, Rickard NS. Emotional Responses to Music: Shifts in Frontal Brain Asymmetry Mark Periods of Musical Change. Front Psychol. 2017 Dec 4;8:2044. doi: 10.3389/fpsyg.2017.02044. eCollection 2017. PMID 29255434